CLINICAL TRIAL: NCT01942720
Title: Monitoring Disease Activity Using Video Capsule Endoscopy (VCE) in Crohn's Disease (CD) Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MA-209
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2016-08

CONDITIONS: Known Crohn Disease Subjects
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capsule endoscopy (Other)
  Interventions: Device: Capsule endoscopy and Ileocolonoscopy tests

INTERVENTIONS:
Device: Capsule endoscopy and Ileocolonoscopy tests

SUMMARY:
This study is designed to evaluate the performance of VCE in the assessment of mucosal inflammation 6 months after the first VCE procedure

DETAILED DESCRIPTION:
This is a prospective, multi-center (up to 15 sites) study which aims to assess the ability of VCE (Video capsule endoscopy) to detect change in the severity of the small bowel mucosal disease activity in CD subjects after 6 months .

Up to 75 subjects will participate in this study. An interim analysis will be done after study completion with 20 subjects. All subjects to be enrolled in this study will be pediatric and\or adult subjects with known Crohn's disease

ELIGIBILITY:
Inclusion Criteria:

1. Subject ages 2-75 years, inclusive
2. Subjects with a diagnosis of known Crohn disease
3. Referred to ileocolonoscopy (up to 4 weeks before the CE procedure)
4. Proven patency by the Agile capsule or another approach deemed clinically acceptable by the investigator, e.g. CT enterography, MRE (Magenetic Resonance Enteroscopy), performed within the 90 days prior to enrollment.
5. Subject or parent agrees to sign consent form

Exclusion Criteria:

The presence of any of the following will exclude a subject from study enrollment:

1. Subjects with change in IBD (Inflammatory Bowel Disease) drug therapy between the baseline ileocolonoscopy and VCE
2. Subjects with a history of prior ileocecectomy, Ileal Pouch-Anal Anastomosis (IPAA) and J pouch or an ostomy
3. Stricture seen on radiological exam.
4. Indeterminate Colitis
5. Ulcerative Colitis
6. Antibiotic Associated Colitis
7. Known history of intestinal obstruction or current obstructive symptoms, such as severe abdominal pain with accompanying nausea or vomiting, based on investigator judgment.
8. Non-steroidal anti-inflammatory drugs including aspirin (twice weekly or more), not including aspirin up to 81mg daily, during the 4 weeks preceding enrollment
9. Suspected GI stricture, followed by PillCam® Patency study or other imaging study that could not prove patency of the GI tract.
10. Subject is expected to undergo MRI examination within 7 days after ingestion of the capsule.
11. Subjects with known or suspected delayed gastric emptying
12. Subjects with known or suspected delayed Small bowel motility
13. Subject has any allergy or other known contraindication to the medications used in the study.
14. Women who are either pregnant or nursing at the time of screening, or are of child-bearing potential and do not agree to practice medically acceptable methods of contraception.
15. Unwillingness to use a medically accepted method of contraception throughout duration of study
16. Concurrent participation in another clinical trial using any investigational drug or device.
17. Subject has cardiac pacemaker or other implanted electromedical devices
18. Subject suffers from a life threatening condition.
19. Subject with a history or clinical evidence of renal disease and/or previous clinically significant laboratory abnormalities of renal function parameters.
20. Subject suffers from any condition, such as swallowing problems, which precludes compliance with study and/or device instructions.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leighton, MD, Principal Investigator — Mayo Clinic; Gil Melmed, MD, Principal Investigator — Cyder Cinai LA
Locations (15):
- United States (15):
  - Mayo Clinic, Scottsdale, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Borland-Groover Clinic, Jacksonville, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Children's Center for Digestive Healthcare, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Indiana Unveresity Hospital, Indianapolis, Indiana
  - Iowa Digestive Disease Center, Clive, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Metropolitan Gastroenterology Group, Chevy Chase, Maryland
  - Digestive Health Center of Michigan, Michigan, Michigan
  - Atlantic Health System Morristown Memorial Pediatric GE, Morristown, New Jersey
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Dr. Romeo, Dayton Gastroenterology, Dayton, Ohio
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia

REFERENCES:
- [Derived] Melmed GY, Dubinsky MC, Rubin DT, Fleisher M, Pasha SF, Sakuraba A, Tiongco F, Shafran I, Fernandez-Urien I, Rosa B, Papageorgiou NP, Leighton JA. Utility of video capsule endoscopy for longitudinal monitoring of Crohn's disease activity in the small bowel: a prospective study. Gastrointest Endosc. 2018 Dec;88(6):947-955.e2. doi: 10.1016/j.gie.2018.07.035. Epub 2018 Aug 4. PMID 30086261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment started on September 2013 and ended on July 2016 74 subjects enrolled within 15 sites in the US
Groups:
- Capsule Endoscopy: Capsule endoscopy and Ileocolonoscopy tests
Period: Overall Study
Arm/Group | Capsule Endoscopy
Started | 74
Completed | 53
Not Completed | 21

BASELINE CHARACTERISTICS:
Arm/Group | Capsule Endoscopy
Number analyzed (Participants) | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 68
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 30
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 74

OUTCOME MEASURES:

1. Primary Outcome: Mucosal Change in VCE (Video Capsule Endoscopy) Mucosal Scores and PGA (Physician Global Assessment)
Description: To correlate the mucosal change in VCE mucosal score (Lewis score and CECDEIS( Capsule Endoscopy Crohn's Disease Endoscopic Index)) with change in Physician Global Assessment of CD activity 6 months after the first VCE procedure; PGA scale: 0-Normal, 1-Mild disease, 2- Moderate Disease, 3-Severe Disease Lewis Score scale: continuance scale variable, higher score higher disease severity (0- unlimited) remission <135 CECDEIS score scale: continuance scale variable, higher score higher disease severity (0-44) , no "normal range" Studies discuss a drop in the number as indicating healing but not a specific cutoff
Time Frame: 6 months changefrom Baseline
Population: Correlation between changes in VCE mucosal scores (Lewis and CECDEIS) and change in PGA score of CD (Crohn's Disease) activity from baseline to follow-up at 6 months; number of participants for this outcome measure includes participants with available data for PGA, SB (small bowel) Lewis score, SB CECDEIS score, respectively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsule Endoscopy
Number analyzed (Participants) | 54
units on a scale
  PGA score change | -0.3 (0.77)
  Total SB Lewis score: number analyzed (Participants) | 49
  Total SB Lewis score | -382.9 (1232.8)
  Total SB CECDEIS score change: number analyzed (Participants) | 49
  Total SB CECDEIS score change | -2.7 (9.05)
Statistical Analysis 1: Comparison: Capsule Endoscopy; Relationship of total PillCam SB Lewis score with PGA score change from baseline visit to 6 month follow-up; Test type: Superiority or Other; p = 0.631, Sperman test; Sperman correlation coeficient = -0.70
Statistical Analysis 2: Comparison: Capsule Endoscopy; Relationship of total PillCam SB CECDEIS score with PGA score change from baseline visit to 6 month follow-up; Test type: Superiority or Other; p = 0.882, Sperman correlation; Sperman correlation coeficient = 0.022

2. Secondary Outcome: Correlation Between SES CD (Simple Endoscopic Score for Chron's Disease) Score and Capsule Scoring Indexes
Description: Evaluate the correlation between SES CD score and capsule scoring indexes (Lewis and CECDEIS) in the TI (Terminal Ileum) at baseline.
  SES CD score scale 0-12, Higher score=higher disease severity Lewis Score scale: continuance scale variable, higher score higher disease severity (0- unlimited) remission <135 CECDEIS score scale: continuance scale variable, higher score higher disease severity (0-44) , no "normal range" Studies discuss a drop in the number as indicating healing but not a specific
Time Frame: Baseline
Population: number of participants for this outcome measure includes participants with available data for SES CD, TI Lewis score, TI CECDEIS score, respectively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsule Endoscopy
Number analyzed (Participants) | 52
units on a scale
  TI SES-CD score at baseline visit | 3.2 (3.62)
  TI Lewis score at baseline | 11941.1 (1874.7)
  TI CECDEIS score at baseline | 14 (15.51)
Statistical Analysis 1: Comparison: Capsule Endoscopy; Relationship of PillCam SB TI Lewis scores with TI SES-CD score at baseline visit; Test type: Superiority or Other; p < 0.001, Sperman correlation; Sperman correlation coefficient = 0.735
Statistical Analysis 2: Comparison: Capsule Endoscopy; Relationship of PillCam SB TI CECDEIS scores with TI SES-CD score at baseline visit; Test type: Superiority or Other; p < 0.001, Sperman correlation; Sperman correlation coefficient = 0.726

3. Secondary Outcome: Correlation Between the Change in SES CD Score and the Change in Capsule Scoring Indexes- in Terminal Ileum
Description: Evaluate the correlation between the change in SES CD score and the change in capsule scoring indexes (Lewis and CECDEIS) in the TI after 6 months SES CD score scale 0-12, Higher score=higher disease severity Lewis Score scale: continuance scale variable, higher score higher disease severity (0- unlimited) remission <135 CECDEIS score scale: continuance scale variable, higher score higher disease severity (0-44) , no "normal range" Studies discuss a drop in the number as indicating healing but not a specific cutoff
Time Frame: 6 months change from Baseline
Population: number of subjects with Colonoscopy score is lower than number of subjects analyzed due to colonoscopy video malfunction. number of participants for this outcome measure includes participants with available data for TI SES CD, TI Lewis, TI CECDEIS scores, respectively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsule Endoscopy
Number analyzed (Participants) | 45
units on a scale
  TI SES-CD score change: number analyzed (Participants) | 40
  TI SES-CD score change | -0.4 (2.88)
  TI Lewis score change | -410.8 (1266.9)
  TI CECDEIS score change | -3.1 (11.55)
Statistical Analysis 1: Comparison: Capsule Endoscopy; Relationship of PillCam SB Lewis score with TI SES-CD score change from baseline visit to 6 month follow-up; Test type: Superiority or Other; p = 0.002, Sperman correlation; Sperman correlation coefficient = 0.493
Statistical Analysis 2: Comparison: Capsule Endoscopy; Relationship of PillCam SB CECDEIS score with TI SES-CD score change from baseline visit to 6 month follow-up; Test type: Superiority or Other; p < 0.001, Sperman correlation; Sperman correlation coefficient = 0.531

4. Secondary Outcome: Evaluate the Entire SB CE Scores
Description: Evaluate the entire SB CE Scores (Lewis & CECDEIS) change as compared to the change at TI in CE Scores (Lewis & CECDEIS).
  Lewis Score scale: continuance scale variable, higher score higher disease severity (0- unlimited) remission <135 CECDEIS score scale: continuance scale variable, higher score higher disease severity (0-44) , no "normal range" Studies discuss a drop in the number as indicating healing but not a specific
Time Frame: 6 months change from Baseline
Population: number of Lewis & CECDEIS TI score change is lower due to inability to identify TI. number of participants for this outcome measure includes participants with available data for total SB Lewis score change, TI Lewis score change, Total CECDEIS score change, TI Lewis score change, respectively
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Capsule Endoscopy
Number analyzed (Participants) | 49
units on a scale
  total SB Lewis score change | -382.9 (1232.8)
  TI Lewis score change: number analyzed (Participants) | 45
  TI Lewis score change | -410.8 (1266.9)
  Total SB CECDEIS score change | -2.7 (9.05)
  TI CECDEIS score change: number analyzed (Participants) | 45
  TI CECDEIS score change | -3.1 (11.55)
Statistical Analysis 1: Comparison: Capsule Endoscopy; Relationship of PillCam total SB Lewis score change with TI Leis score change from baseline visit to 6 month follow-up; Test type: Superiority or Other; p < 0.001, Sperman correlation; Sperman correlation coefficient = 0.752
Statistical Analysis 2: Comparison: Capsule Endoscopy; Relationship of PillCam total SB CECDEIS score change with TI Leis score change from baseline visit to 6 month follow-up; Test type: Superiority or Other; p < 0.001, Sperman correlation; Sperman correlation coefficient = 0.785

5. Secondary Outcome: Adverse Events (AE)
Description: To assess safety related to capsule retention and other adverse events
Time Frame: 6 months
Population: all enrolled subjects
Measure: Number; unit: AE incidents
Arm/Group | Capsule Endoscopy
Number analyzed (Participants) | 74
AE incidents
  Incidence of Serious Adverse Events | 5
  Incidence of Non-Serious Adverse Events | 59
  Incidence of Anticipated Adverse Events | 0
  Incident of Serious Unanticipated Adverse Events | 5

ADVERSE EVENTS:
Time Frame: Adverse events data collected from subject enrollment up to end of study
Description: all adverse events identified on study subjects were collected from patient enrollment up to end of study duration: AE related and not related to study procedure and or product as well as anticipated and unanticipated AEs
Arm/Group | Capsule Endoscopy
Serious Adverse Events (participants affected / at risk) | 3/74
Other Adverse Events (participants affected / at risk) | 24/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capsule Endoscopy (N=74)
Worsening of IBD, Nausea, vomiting, diarrhea, abdominal pain (Gastrointestinal disorders) | 2 (2) — Unanticipated serious adverse event not related to study device
Asthma Excerbation, Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Unanticipated serious adverse event not related to study device
Pancreatitis, Acute (Hepatobiliary disorders) | 1 (1) — Unanticipated serious adverse event not related to study device
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capsule Endoscopy (N=74)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) — non-serious AE
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) — non-serious AE
Athralgia Of Hands And Elbows, Arthritis Flare (Musculoskeletal and connective tissue disorders) | 2 (2) — non-serious AE
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — non-serious AE
Bilateral Bursitis In Hips (Musculoskeletal and connective tissue disorders) | 1 (1) — non-serious AE
Blolating (Gastrointestinal disorders) | 1 (1) — non-serious AE
Bruise At Venipucture Site. Right Anticubital Space (Injury, poisoning and procedural complications) | 1 (1) — non-serious AE
Bruised Coccyx Due To Fall (Injury, poisoning and procedural complications) | 1 (1) — non-serious AE
C-Difficile (Gastrointestinal disorders) | 1 (1) — non-serious AE
Chest Pain (Cardiac disorders) | 1 (1) — non-serious ae
Common Cold, cough (Infections and infestations) | 2 (2) — non-serious
Crohn's Flare (Gastrointestinal disorders) | 1 (1) — non-serious AE
Cyst Right Great Toe (Injury, poisoning and procedural complications) | 1 (1) — non-serious AE
Detached Retina (Eye disorders) | 1 (1) — non-serious
Diarrhea (Gastrointestinal disorders) | 4 (4) — non-serious
Fatigue (General disorders) | 1 (1) — non-serious
fell (Injury, poisoning and procedural complications) | 1 (1) — non-serious
Flu (Infections and infestations) | 2 (2) — non-serious
Heartburn (Cardiac disorders) | 1 (1) — non-serious AE
Hyponatremia (Injury, poisoning and procedural complications) | 1 (1) — non-serious AE
Incontinence a Little Worse And More Often (Renal and urinary disorders) | 1 (1) — non-serious AE
Iron Deficiency Anemia (Hepatobiliary disorders) | 1 (1) — non-serious AE
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) — non-serious AE
Light Headed (General disorders) | 1 (1) — non-serious AE
Mild Perianal Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — non-serious AE
Nasal congestion (Infections and infestations) | 2 (2) — non-serious AE
Nausea (Gastrointestinal disorders) | 3 (4) — non-serious AE
Pulled Upper Back Muscle Left Side (Musculoskeletal and connective tissue disorders) | 1 (1) — non-serious AE
Questionable Right Lower Quadrant Mass (General disorders) | 1 (1) — non-serious AE
Rash (Skin and subcutaneous tissue disorders) | 4 (4) — non-serious AE
Rectal Urgency (Gastrointestinal disorders) | 1 (1) — non-serious AE
Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — non-serious AE
Right Leg Bruising Secondary To Fall (Injury, poisoning and procedural complications) | 1 (1) — non-serious AE
Strep Throat (Infections and infestations) | 1 (1) — non-serious AE
Superficial Blood Clot Left Axilla Area (General disorders) | 1 (1) — non-serious AE
Syncope (General disorders) | 1 (1) — non-serious AE
Vomiting (Gastrointestinal disorders) | 6 (6) — non-serious AE
Worsening Diabetes (Metabolism and nutrition disorders) | 1 (1) — non-serious AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No